CLINICAL TRIAL: NCT03260322
Title: A Phase 1b Study of ASP8374, an Immune Checkpoint Inhibitor, as a Single Agent and in Combination With Pembrolizumab in Subjects With Advanced Solid Tumors
Brief Title: A Multiple-dose Study of ASP8374, an Immune Checkpoint Inhibitor, as a Single Agent and in Combination With Pembrolizumab in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8374-CL-0101; 2018-001146-34 (EudraCT Number); KEYNOTE KN-A72 (Other: Merck)
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumors
Keywords: Pembrolizumab; Oncology; Tumors; ASP8374; Locally advanced or metastatic solid tumor malignancies
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (17):
- ASP8374 0.5 mg - Monotherapy Dose Escalation (Experimental): Participants received ASP8374 0.5 mg intravenously, on day 1 of every 3 week cycle for a period of up to 16 cycles or until a discontinuation criterion was met during treatment period. Qualifying participants entered re-treatment period and received treatment for an additional 16 cycles or until a discontinuation criteria was met.
  Interventions: Drug: ASP8374
- ASP8374 2 mg - Monotherapy Dose Escalation (Experimental): Participants received ASP8374 2 mg intravenously, on day 1 of every 3 week cycle for a period of up to 16 cycles or until a discontinuation criterion was met during treatment period. Qualifying participants entered re-treatment period and received treatment for an additional 16 cycles or until a discontinuation criteria was met.
  Interventions: Drug: ASP8374
- ASP8374 7 mg - Monotherapy Dose Escalation (Experimental): Participants received ASP8374 7 mg intravenously, on day 1 of every 3 week cycle for a period of up to 16 cycles or until a discontinuation criterion was met during treatment period. Qualifying participants entered re-treatment period and received treatment for an additional 16 cycles or until a discontinuation criteria was met.
  Interventions: Drug: ASP8374
- ASP8374 20 mg - Monotherapy Dose Escalation (Experimental): Participants received ASP8374 20 mg intravenously, on day 1 of every 3 week cycle for a period of up to 16 cycles or until a discontinuation criterion was met during treatment period. Qualifying participants entered re-treatment period and received treatment for an additional 16 cycles or until a discontinuation criteria was met.
  Interventions: Drug: ASP8374
- ASP8374 70 mg - Monotherapy Dose Escalation (Experimental): Participants received ASP8374 70 mg intravenously, on day 1 of every 3 week cycle for a period of up to 16 cycles or until a discontinuation criterion was met during treatment period. Qualifying participants entered re-treatment period and received treatment for an additional 16 cycles or until a discontinuation criteria was met.
  Interventions: Drug: ASP8374
- ASP8374 200 mg - Monotherapy Dose Escalation (Experimental): Participants received ASP8374 200 mg intravenously, on day 1 of every 3 week cycle for a period of up to 16 cycles or until a discontinuation criterion was met during treatment period. Qualifying participants entered re-treatment period and received treatment for an additional 16 cycles or until a discontinuation criteria was met.
  Interventions: Drug: ASP8374
- ASP8374 700 mg - Monotherapy Dose Escalation (Experimental): Participants received ASP8374 700 mg intravenously, on day 1 of every 3 week cycle for a period of up to 16 cycles or until a discontinuation criterion was met during treatment period. Qualifying participants entered re-treatment period and received treatment for an additional 16 cycles or until a discontinuation criteria was met.
  Interventions: Drug: ASP8374
- ASP8374 1400 mg - Monotherapy Dose Escalation (Experimental): Participants received ASP8374 1400 mg intravenously, on day 1 of every 3 week cycle for a period of up to 16 cycles or until a discontinuation criterion was met during treatment period. Qualifying participants entered re-treatment period and received treatment for an additional 16 cycles or until a discontinuation criteria was met.
  Interventions: Drug: ASP8374
- ASP8374 1400 mg - Monotherapy Dose Expansion (Experimental): Participant received ASP8374 1400 mg intravenously, on day 1 of every 3 week cycle for a period of up to 16 cycles or until a discontinuation criterion was met during treatment period. Qualifying participants entered re-treatment period and received treatment for an additional 16 cycles or until a discontinuation criteria was met.
  Interventions: Drug: ASP8374
- ASP8374 20 mg - Combination Dose Escalation (Experimental): Participants received ASP8374 20 mg intravenously in combination with pembrolizumab 200 mg adminstered as a 30 minutes intravenous infusion, on day 1 of every 3 week cycle for a period of up to 16 cycles or until a discontinuation criterion was met. Qualifying participants received combination treatment for an additional 16 cycles or until a discontinuation criteria was met. Participants who completed 16 cycles of combination treatment who entered the follow-up period with PR or SD were allowed to continue on pembrolizumab alone for a period of up to an additional 19 cycles. If the participant was eligible for the re-treatment period during follow up, administration of pembrolizumab alone was discontinued and combination therapy with ASP8374 was resumed per the protocol.
  Interventions: Drug: ASP8374; Drug: Pembrolizumab
- ASP8374 70 mg - Combination Dose Escalation (Experimental): Participants received ASP8374 70 mg intravenously in combination with pembrolizumab 200 mg adminstered as a 30 minutes intravenous infusion, on day 1 of every 3 week cycle for a period of up to 16 cycles or until a discontinuation criterion was met. Qualifying participants received combination treatment for an additional 16 cycles or until a discontinuation criteria was met. Participants who completed 16 cycles of combination treatment who entered the follow-up period with PR or SD were allowed to continue on pembrolizumab alone for a period of up to an additional 19 cycles. If the participant was eligible for the re-treatment period during follow up, administration of pembrolizumab alone was discontinued and combination therapy with ASP8374 was resumed per the protocol.
  Interventions: Drug: ASP8374; Drug: Pembrolizumab
- ASP8374 200 mg - Combination Dose Escalation (Experimental): Participants received ASP8374 200 mg intravenously in combination with pembrolizumab 200 mg adminstered as a 30 minutes intravenous infusion, on day 1 of every 3 week cycle for a period of up to 16 cycles or until a discontinuation criterion was met. Qualifying participants received combination treatment for an additional 16 cycles or until a discontinuation criteria was met. Participants who completed 16 cycles of combination treatment who entered the follow-up period with PR or SD were allowed to continue on pembrolizumab alone for a period of up to an additional 19 cycles. If the participant was eligible for the re-treatment period during follow up, administration of pembrolizumab alone was discontinued and combination therapy with ASP8374 was resumed per the protocol.
  Interventions: Drug: ASP8374; Drug: Pembrolizumab
- ASP8374 700 mg - Combination Dose Escalation (Experimental): Participants received ASP8374 700 mg intravenously in combination with pembrolizumab 200 mg adminstered as a 30 minutes intravenous infusion, on day 1 of every 3 week cycle for a period of up to 16 cycles or until a discontinuation criterion was met. Qualifying participants received combination treatment for an additional 16 cycles or until a discontinuation criteria was met. Participants who completed 16 cycles of combination treatment who entered the follow-up period with PR or SD were allowed to continue on pembrolizumab alone for a period of up to an additional 19 cycles. If the participant was eligible for the re-treatment period during follow up, administration of pembrolizumab alone was discontinued and combination therapy with ASP8374 was resumed per the protocol.
  Interventions: Drug: ASP8374; Drug: Pembrolizumab
- ASP8374 1400 mg - Combination Dose Escalation (Experimental): Participants received ASP8374 1400 mg intravenously in combination with pembrolizumab 200 mg adminstered as a 30 minutes intravenous infusion, on day 1 of every 3 week cycle for a period of up to 16 cycles or until a discontinuation criterion was met. Qualifying participants received combination treatment for an additional 16 cycles or until a discontinuation criteria was met. Participants who completed 16 cycles of combination treatment who entered the follow-up period with PR or SD were allowed to continue on pembrolizumab alone for a period of up to an additional 19 cycles. If the participant was eligible for the re-treatment period during follow up, administration of pembrolizumab alone was discontinued and combination therapy with ASP8374 was resumed per the protocol.
  Interventions: Drug: ASP8374; Drug: Pembrolizumab
- ASP8374 200 mg - Combination Dose Expansion (Experimental): Participants received ASP8374 200 mg intravenously in combination with pembrolizumab 200 mg adminstered as a 30 minutes intravenous infusion, on day 1 of every 3 week cycle for a period of up to 16 cycles or until a discontinuation criterion was met. Qualifying participants received combination treatment for an additional 16 cycles or until a discontinuation criteria was met. Participants who completed 16 cycles of combination treatment who entered the follow-up period with PR or SD were allowed to continue on pembrolizumab alone for a period of up to an additional 19 cycles. If the participant was eligible for the re-treatment period during follow up, administration of pembrolizumab alone was discontinued and combination therapy with ASP8374 was resumed per the protocol.
  Interventions: Drug: ASP8374; Drug: Pembrolizumab
- ASP8374 700 mg - Combination Dose Expansion (Experimental): Participants received ASP8374 700 mg intravenously in combination with pembrolizumab 200 mg adminstered as a 30 minutes intravenous infusion, on day 1 of every 3 week cycle for a period of up to 16 cycles or until a discontinuation criterion was met. Qualifying participants received combination treatment for an additional 16 cycles or until a discontinuation criteria was met. Participants who completed 16 cycles of combination treatment who entered the follow-up period with PR or SD were allowed to continue on pembrolizumab alone for a period of up to an additional 19 cycles. If the participant was eligible for the re-treatment period during follow up, administration of pembrolizumab alone was discontinued and combination therapy with ASP8374 was resumed per the protocol.
  Interventions: Drug: ASP8374; Drug: Pembrolizumab
- ASP8374 1400 mg - Combination Dose Expansion (Experimental): Participants received ASP8374 1400 mg intravenously in combination with pembrolizumab 200 mg adminstered as a 30 minutes intravenous infusion, on day 1 of every 3 week cycle for a period of up to 16 cycles or until a discontinuation criterion was met. Qualifying participants received combination treatment for an additional 16 cycles or until a discontinuation criteria was met. Participants who completed 16 cycles of combination treatment who entered the follow-up period with PR or SD were allowed to continue on pembrolizumab alone for a period of up to an additional 19 cycles. If the participant was eligible for the re-treatment period during follow up, administration of pembrolizumab alone was discontinued and combination therapy with ASP8374 was resumed per the protocol.
  Interventions: Drug: ASP8374; Drug: Pembrolizumab

INTERVENTIONS:
Drug: ASP8374 — intravenous
Drug: Pembrolizumab — intravenous
  Other Names: Keytruda
  Arms: ASP8374 1400 mg - Combination Dose Escalation; ASP8374 1400 mg - Combination Dose Expansion; ASP8374 20 mg - Combination Dose Escalation; ASP8374 200 mg - Combination Dose Escalation; ASP8374 200 mg - Combination Dose Expansion; ASP8374 70 mg - Combination Dose Escalation; ASP8374 700 mg - Combination Dose Escalation; ASP8374 700 mg - Combination Dose Expansion

SUMMARY:
The primary purpose of this study is to evaluate the tolerability and safety profile of ASP8374 when administered as a single agent and in combination with pembrolizumab in participants with locally advanced (unresectable) or metastatic solid tumor malignancies. Also primary purpose is to characterize the pharmacokinetic profile of ASP8374 when administered as a single agent and in combination with pembrolizumab. Last primary purpose of this study is to determine the recommended Phase 2 dose (RP2D) of ASP8374 when administered as a single agent and in combination with pembrolizumab.

The secondary purpose of this study is to evaluate the anti-tumor effect (objective response rate [ORR], duration of response [DOR], persistence of response after discontinuation, and disease control rate [DCR]) of ASP8374 when administered as a single agent and in combination with pembrolizumab.

NTP: Neutropenia

NHAE:Non-haematological AE

GBS: Guillain-Barré syndrome""

IRR: Infusion-related reaction

AST: Aspartate aminotransferase

ALT: Alanine aminotransferase

MS/MG: Myasthenia Syndrome/Myasthenia Gravis

TRT: Treatment-related Toxicity

TCP: Thrombocytopenia

DETAILED DESCRIPTION:
This is a multi-center, multiple-dose, dose-escalation and expansion study of ASP8374 as a single agent and in combination with pembrolizumab. After discontinuation of study drug treatment (initial treatment and re-treatment), all participants will complete an end of treatment visit along with 30-day and 90-day safety follow-up visits from the last dose of ASP8374. Participants will be enrolled in respectively escalation cohorts or expansion cohorts. The 90-day safety follow-up visit is optional for participants who discontinue due to progressive disease or initiate new anticancer treatment after the last dose of study drug.

Escalation cohorts: Approximately 60 participants may be enrolled in the escalation cohorts (approximately 30 participants for monotherapy and 30 participants for combination therapy).

Expansion cohorts: The total number of subjects in the expansion cohorts will depend on the observed pharmacokinetic and antitumor activity. It is estimated that approximately 240 participants may be enrolled in the monotherapy and combination therapy expansion cohorts.

As the number of participants in the escalation cohorts and the expansion cohorts will depend on the observed Dose Limiting Toxicity (DLT), pharmacokinetics and antitumor activity, approximately 300 participants are expected to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Subject has locally-advanced (unresectable) or metastatic solid tumor malignancy (no limit to the number of prior treatment regimens) that is confirmed by available pathology records or current biopsy as well as:

  * Subject in the escalation cohort has received all standard therapies (unless the therapy is contraindicated or intolerable) felt to provide clinical benefit for the subject's specific tumor type. OR
  * Subject in an expansion cohort has received at least one standard therapy for the subject's specific tumor type.
* For Korea, Italy and Portugal only: Subject has locally-advanced (unresectable) or metastatic solid tumor malignancy (no limit to the number of prior treatment regimens) that is confirmed by available pathology records or current biopsy and has received all standard therapies (unless the therapy is contraindicated or intolerable) felt to provide clinical benefit for the subject's specific tumor type.
* Subject has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2.
* Subject's last dose of prior antineoplastic therapy, including any immunotherapy, was 21 days or 5 half-lives, whichever is shorter, prior to initiation of study drug administration. A subject with epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) mutation-positive NSCLC is allowed to remain on EGFR tyrosine kinase inhibitor (TKI) therapy or ALK inhibitor until 4 days prior to the start of study drug administration.
* For Korea only: Subject's last dose of prior antineoplastic therapy, including any immunotherapy, was at least 21 days or 5 half-lives, whichever is shorter, prior to initiation of study drug administration. For drugs with a half-life greater than or equal to 21 days, the investigator should consider if this washout is sufficient. A subject with epidermal growth factor receptor (EGFR) mutation-positive non-small cell lung cancer (NSCLC) is allowed to remain on EGFR tyrosine kinase inhibitor (TKI) therapy until 7 days prior to the start of study drug administration.
* Subject has completed any radiotherapy (including stereotactic radiosurgery) at least 2 weeks prior to study drug administration.
* Subject's adverse events (excluding alopecia) from prior therapy have improved to grade 1 or baseline within 14 days prior to start of study treatment.
* Subject with metastatic castration resistant prostate cancer (mCRPC) (positive bone scan and/or soft tissue disease documented by computed tomography (CT) / magnetic resonance imaging (MRI)) meets both of the following:

  * Subject has serum testosterone ≤ 50 ng/dL at screening.
  * Subject has had an orchiectomy or plans to continue androgen deprivation therapy (ADT) for the duration of study treatment.
* Subject has adequate organ function prior to start of study treatment as indicated by the following laboratory values. If a subject has received a recent blood transfusion, the laboratory tests must be obtained ≥ 4 weeks after any blood transfusion.
* Female subject is eligible to participate if she is not pregnant and at least 1 of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance throughout the treatment period and for at least 6 months after the final study drug administration.
* Female subject must agree not to breastfeed starting at screening and throughout the study treatment, and for 6 months after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study treatment, and for 6 months after the final study drug administration.
* A male subject with female partner(s) of childbearing potential must agree to use contraception as detailed during the treatment period and for at least 6 months after the final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study treatment, and for 6 months after the final study drug administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the study treatment and for 6 months after the final study drug administration.
* Subject agrees not to participate in another interventional study while receiving study drug (subjects who are currently in the follow-up period of an interventional clinical trial are allowed).

Additional Inclusion Criteria for Subjects in the Expansion Cohorts:

* Subject meets one of the following:

  * Subject has the tumor type for which a confirmed response was observed in a monotherapy or combination therapy dose escalation cohort; or
  * For an expansion cohort opened due to achieving predicted efficacious exposure, subject has squamous cell carcinoma of the head and neck (SCCHN); or
  * For tumor specific expansion cohorts of ASP8374 with pembrolizumab, subject has the applicable tumor type (e.g., non-small cell lung cancer (NSCLC), bladder cancer, gastric cancer, metastatic castration resistant prostate cancer (MCRPC) or colorectal cancer (CRC)).
* Subject has at least 1 measureable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions. Subjects with mCRPC who do not have measurable lesions must have at least one of the following:

  * Progression with 2 or more new bone lesions; or
  * Prostate-specific antigen (PSA) progression (defined as a minimum of three rising PSA levels with an interval of ≥ 1 week between each determination) within 6 weeks prior to study drug administration and a PSA value at the screening visit ≥ 2 ng/mL.
* Subject consents to provide an available tumor specimen in a tissue block or unstained serial slides obtained within 56 days prior to first dose of study treatment, or subject is an appropriate candidate for tumor biopsy and is amenable to undergoing a tumor biopsy (core needle biopsy or excision) during the screening period.This does not apply to subjects with mCRPC without measurable disease.
* Subject in any expansion cohort, is an appropriate candidate for tumor biopsy and consents to undergoing a tumor biopsy (core needle biopsy or excision) during the treatment period as indicated in the Schedule of Assessments.

Exclusion:

* Subject weighs < 45 kg at screening.
* Subject has received investigational therapy (other than an investigational epidermal growth factor receptor tyrosine kinase inhibitor (EGFR TKI) in a subject with EGFR activating mutations or ALK inhibitor in a subject with an ALK mutation) within 21 days or 5 half-lives, whichever is shorter, prior to start of study drug.
* Subject requires or has received systemic steroid therapy or any other immunosuppressive therapy within 14 days prior to study drug administration. Subjects using a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 30 mg per day of hydrocortisone up to 10 mg per day of prednisone) are allowed.
* Subject has symptomatic central nervous system (CNS) metastases or subject has evidence of unstable CNS metastases even if asymptomatic (e.g., progression on scans). Subjects with previously treated CNS metastases are eligible, if subject is clinically stable and have no evidence of CNS progression by imaging for at least 4 weeks prior to start of study treatment and are not requiring immunosuppressive doses of systemic steroids (> 30 mg per day of hydrocortisone or > 10 mg per day of prednisone or equivalent) for longer than 2 weeks.
* Subject has an active autoimmune disease. Subjects with type 1 diabetes mellitus, endocrinopathies stably maintained on appropriate replacement therapy, or skin disorders (e.g., vitiligo, psoriasis, or alopecia) not requiring systemic treatment are allowed.
* Subject was discontinued from prior immunomodulatory therapy due to a grade ≥ 3 toxicity that was mechanistically related (e.g., immune related) to the agent.
* Subject has known history of serious hypersensitivity reaction to a known ingredient of ASP8374 or pembrolizumab or severe hypersensitivity reaction to treatment with another monoclonal antibody.
* Subject has a known history of Human Immunodeficiency Virus.
* Subject with positive for Hepatitis B virus (HBV) antibodies and surface antigen (including acute HBV or chronic HBV) or Hepatitis C ([HCV]; ribonucleic acid [RNA] detected by qualitative assay). Hepatitis C RNA testing is not required in subjects with negative Hepatitis C antibody testing.
* Subject has received a live vaccine against infectious diseases within 28 days prior to initiation of study treatment.
* Subject has a history of drug-induced pneumonitis (interstitial lung disease), a history of (non-infectious) pneumonitis that required steroids, radiation pneumonitis or currently has pneumonitis.
* Subject has an infection requiring systemic therapy within 14 days prior to study drug treatment.
* Subject has received a prior allogeneic bone marrow or solid organ transplant.
* Subject is expected to require another form of antineoplastic therapy while on study treatment.
* Subject has had a myocardial infarction or unstable angina within 6 months prior to the start of study treatment or currently has an uncontrolled illness including, but not limited to symptomatic congestive heart failure, clinically significant cardiac disease, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Any condition that makes the subject unsuitable for study participation.
* Subject has had a major surgical procedure and has not completely recovered within 28 days prior to the start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) | Up to 21 Days (For ASP8374 0.5 mg: Up to 7 days)
  DLT was defined as any of the following AE that cannot clearly attribute to a cause other than study drug:
  Grade (Gr) 4 NTP or Gr ≥ 3 febrile NTP Gr 4 TCP; or Gr 3 TCP accompanied by bleeding that required any transfusion Gr 4 anemia or Gr 3 anemia requiring transfusion Gr ≥ 3 NHAE Gr ≥ 2 pneumonitis Gr ≥ 2 encephalopathy, meningitis, or motor or sensory neuropathy AST or ALT > 5x upper limit of normal (ULN; Gr ≥ 3) without liver metastases AST or ALT > 8 x ULN in participants with liver metastases AST or ALT > 3 x ULN & total bilirubin > 2 x ULN (in participant with Gilbert syndrome: AST or ALT > 3x ULN & direct bilirubin > 1.5 x ULN) Total bilirubin > 3x ULN (Gr ≥ 3) GBS or MS/MG IRR that required the infusion to be discontinued Prolonged delay (> 2 weeks) in initiating cycle 2 due to TRT Any TRT that caused the participant to discontinue treatment during cycle 1 Missing >25% of ASP8374 or pembrolizumab doses as a result of drug-related AE(s) during the 1st cycle Gr 5 toxicity
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | From first dose up to 90 days after last dose (maximum duration: 938 days)
  An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An AE is considered "serious" if, it results in any of the following outcomes:
  results in death; is life-threatening; results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions; results in congenital anomaly, or birth defect; requires inpatient hospitalization; or leads to prolongation of hospitalization; other medically important events. TEAE was defined as an AE observed after starting administration of the study drug.
Number of Participants with Infusion Related Reactions | From first dose up to 90 days after last dose (maximum duration: 938 days)
  Number of participants with infusion related reactions are reported.
Number of Participants with Immune- Related Treatment Emergent Adverse Events (IrTEAEs) | From first dose up to 90 days after last dose (maximum duration: 938 days)
  AEs associated with pembrolizumab exposure may represent an immune-related response. Immune-related AEs observed with currently approved check point inhibitor CPIs include rash, oral mucositis, dry mouth, colitis/diarrhea, hepatitis, pneumonitis, and endocrinopathies (hypophysitis, hypothyroidism, hyperthyroidism, adrenal insufficiency and Type 1 diabetes mellitus). Other less frequent irAEs associated with CPIs include: nephritis; pancreatitis; myositis; arthritis; neurologic toxicities (Guillain-Barre syndrome, myasthenia gravis, posterior reversible encephalopathy syndrome, aseptic meningitis, enteric neuropathy, transverse myelitis, and autoimmune encephalitis), cardiotoxicity (myocarditis and conduction abnormalities); hematologic toxicity (red cell aplasia, neutropenia, thrombo-cytopenia, acquired hemophilia A, and cryoglobulinemia); and eye inflammation (episcleritis, conjunctivitis, uveitis or orbital inflammation).
Number of Participants with Eastern Cooperative Oncology Group (ECOG) Performance status | End of treatment ASP8374 (Up to 427 days)
  The ECOG was used to assess performance status. Number of participants in each of the ECOG PS grade were reported.
  0 = Fully active, able to carry on all predisease performance without restriction;
  1. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature;
  2. Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours;
  3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours;
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
Pharmakokinetics (PK) of ASP8374 (Cycle 1): Area Under the Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUClast) (Monotherapy Dose Escalation Cohort) | Cycles 1: predose, end of dosing (within 20 minutes), 4hr, 24hr, 48hr, 168hr, 336hr postdose (each cycle = 21 days)
  Area under the concentration-time curve from the time zero to the last measurable concentration was derived from the plasma samples.
Pharmakokinetics (PK) of ASP8374 (Cycle 7): Area Under the Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUClast) (Monotherapy Dose Escalation Cohort) | Cycles 7: predose, end of dosing (within 20 minutes), 4hr, 24hr, 48hr, 168hr, 336hr postdose (each cycle = 21 days)
  Area under the concentration-time curve from the time zero to the last measurable concentration was derived from the plasma samples.
PK of ASP8374 (Cycle 1): Area Under the Concentration-Time Curve From the Time of Dosing Extrapolated to Time Infinity (AUCinf) (Monotherapy Dose Escalation Cohort) | Cycle 1: predose. end of dosing, 4hr, 24hr, 48hr, 168hr, 336hr postdose (each cycle = 21 days)
  Area under the concentration-time curve from the time of dosing extrapolated to time infinity was derived from the plasma samples.
PK of ASP8374 (Cycle 1): Percentage of AUCinf due to extrapolation from the last measurable concentration to time infinity [AUCinf(%extrap)] (Monotherapy Dose Escalation Cohort) | Cycle 1: predose. end of dosing, 4hr, 24hr, 48hr, 168hr, 336hr postdose (each cycle = 21 days)
  Percentage of AUCinf due to extrapolation from the last measurable concentration to time infinity was derived from the plasma samples.
PK of ASP8374 (Cycle 7): Area Under the Concentration-Time Curve From the Time of Dosing to the Start of the Next Dosing Interval at Multiple Dose Conditions (AUCtau) (Monotherapy Dose Escalation Cohort) | Cycle 7: predose. end of dosing, 4hr, 24hr, 48hr, 168hr, 336hr postdose (each cycle= 21 days)
  AUCtau: Area under the concentration-time curve from the time of dosing to the start of the next dosing interval was derived from plasma samples.
PK of ASP8374 (Cycle 1): Maximum Plasma concentration (Cmax) (Monotherapy Dose Escalation Cohort) | Cycles 1: predose, end of dosing (within 20 minutes), 4hr, 24hr, 48hr, 168hr, 336hr postdose (each cycle = 21 days)
  Maximum plasma concentration of ASP8374 was derived from the plasma samples.
PK of ASP8374 (Cycle 7): Cmax (Monotherapy Dose Escalation Cohort) | Cycles 7: predose, end of dosing (within 20 minutes), 4hr, 24hr, 48hr, 168hr, 336hr postdose (each cycle = 21 days)
  Maximum plasma concentration of ASP8374 was derived from the plasma samples.
PK of ASP8374 (Cycle 7): Trough concentration (Ctrough) (Monotherapy Dose Escalation Cohort) | Cycle 7: predose
  Trough Concentration was derived from the PK samples.
PK of ASP8374 (Cycle 1): Time of Maximum Concentration (Tmax) (Monotherapy Dose Escalation Cohort) | Cycles 1: predose, end of dosing (within 20 minutes), 4hr, 24hr, 48hr, 168hr, 336hr postdose (each cycle = 21 days)
  Time of maximum plasma concentration of ASP8374 was derived from the plasma samples.
PK of ASP8374 (Cycle 7): Tmax (Monotherapy Dose Escalation Cohort) | Cycles 7: predose, end of dosing (within 20 minutes), 4hr, 24hr, 48hr, 168hr, 336hr postdose (each cycle = 21 days)
  Time of maximum plasma concentration of ASP8374 was derived from the plasma samples.
PK of ASP8374 (Cycle 1): Terminal Elimination Half-life (T1/2) of ASP8374 (Monotherapy Dose Escalation Cohort) | Cycle 1: predose. end of dosing, 4hr, 24hr, 48hr, 168hr, 336hr postdose (each cycle = 21 days)
  Terminal half life of ASP8374 was derived from the plasma samples.
PK of ASP8374 (Cycle 1): Time of Last Measurable Concentration (tlast) (Monotherapy Dose Escalation Cohort) | Cycles 1: predose, end of dosing (within 20 minutes), 4hr, 24hr, 48hr, 168hr, 336hr postdose (each cycle = 21 days)
  Time of last measurable concentration was derived from the plasma samples.
PK of ASP8374 (Cycle 7): tlast (Monotherapy Dose Escalation Cohort) | Cycles 7: predose, end of dosing (within 20 minutes), 4hr, 24hr, 48hr, 168hr, 336hr postdose (each cycle = 21 days)
  Time of last measurable concentration was derived from the plasma samples.
PK of ASP8374 (Cycle 1): Total Systemic Observed Clearance After Intravenous Dosing (CLobs) of ASP8374 (Monotherapy Dose Escalation Cohort) | Cycles 1: predose, end of dosing (within 20 minutes), 4hr, 24hrt, 48hr, 168hr, 336hr postdose (each cycle = 21 days)
  Total systemic observed clearance after intravenous dosing was derived from the plasma samples
PK of ASP8374 (Cycle 1): Volume of Distribution During the Terminal Elimination Phase (Vz) after Intravenous Dosing (Monotherapy Dose Escalation Cohort) | Cycle 1: predose. end of dosing, 4hr, 24hr, 48hr, 168hr, 336hr postdose (each cycle = 21 days)
  Volume of distribution after intravenous dosing during the terminal elimination phase was derived from plasma samples.
PK of ASP8374 (Cycle 7): Apparent Volume of Distribution at Steady State (Vss) after Intravenous Dosing of ASP8374 (Monotherapy Dose Escalation Cohort) | Cycle 7: predose. end of dosing, 4hr, 24hr, 48hr, 168hr, 336hr postdose (each cycle= 21 days)
  Volume of distribution at steady state after intravenous dosing was derived from plasma samples.

SECONDARY OUTCOMES:
Best Overall Response (BOR) as per RECIST as per Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1) | From start of study until radiographical progression or date of censoring (maximum duration: 938 days)
  The BOR rate was defined as the percentage of participants whose best response was Complete Response (CR) or Partial Response (PR) as defined by RECIST v1.1 criteria. CR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. PR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters.
BOR as per immune Response Evaluation Criteria in Solid Tumors (iRECIST) | From start of study until radiographical progression or date of censoring (maximum duration: 938 days)
  The BOR rate was defined as the percentage of participants whose best response was immune complete response (iCR) or immune partial response (iPR) as defined by RECIST v1.1 criteria. immune complete response (iCR) or immune partial response (iPR). iCR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. iPR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters.
Objective Response Rate (ORR) as per RECIST v1.1 | From start of study until radiographical progression or date of censoring (maximum duration: 938 days)
  ORR as per RECIST v1.1 was defined as the percentage of participants for each dose level whose best overall response was rated as confirmed CR or PR. CR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. PR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters.
ORR as per iRECIST | From start of study until radiographical progression or date of censoring (maximum duration: 938 days)
  ORR as per iRECIST was defined as the percentage of participants for each dose level whose best overall response was rated as confirmed iCR or iPR. iCR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. iPR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters.
Duration of Response as per RECIST v1.1 | From the date of the first response CR/PR to the date of radiographical progression or date of censoring (maximum 938 days)
  DOR as per RECIST v1.1 was defined as the time from the date of the first response CR/PR (whichever is first recorded) to the date of radiographical progression or date of censoring. CR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. PR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters.
DOR as per iRECIST | From the date of the first response iCR/iPR to the date of radiographical progression or date of censoring (maximum 938 days)
  DOR as per iRECIST was defined as the time from the date of the first response iCR/iPR (whichever is first recorded) to the date of radiographical progression or date of censoring. iCR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. iPR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters.
Persistence of Response After Discontinuation as per RECIST v1.1 | From date of treatment discontinuation to the date of radiographical progression or date of censoring (maximum duration: 938 days)
  Persistence of response as per RECIST v1.1 was defined as the time from the date of treatment discontinuation to the date of radiographical progression or date of censoring. Persistence of response was derived for participants who at the time of treatment discontinuation had a confirmed response of CR or PR based on RECIST 1.1. CR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. PR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters.
Persistence of Response After Discontinuation as per iRECIST | From date of treatment discontinuation to the date of radiographical progression or date of censoring (maximum duration: 938 days)
  Persistence of response as per iRECIST was defined as the time from the date of treatment discontinuation to the date of radiographical progression or date of censoring. Persistence of response was derived for participants who at the time of treatment discontinuation had a confirmed response of iCR or iPR. iCR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. iPR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters.
Disease Control Rate (DCR) as per RECIST v1.1 | From start of study until radiographical progression or date of censoring (maximum duration: 938 days)
  DCR as per RECIST v1.1 was defined as the percentage of participants for each dose level whose best overall response is rated as confirmed CR, PR or Stable Disease (SD). CR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. PR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters. SD was defined as neither sufficient decrease to qualify for PR nor sufficient increase to qualify for progressive disease taking as reference the smallest sum of diameters.
Disease Control Rate (DCR) as per iRECIST | From start of study until radiographical progression or date of censoring (maximum duration: 938 days)
  DCR as per iRECIST was defined as the perccentage of participants for each dose level whose best overall response is rated as confirmed iCR, iPR or immune Stable Disease (iSD). iCR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. iPR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters. iSD was defined as neither sufficient decrease to qualify for PR nor sufficient increase to qualify for progressive disease taking as reference the smallest sum of diameters.
Time to Response as per RECIST v1.1 | From first dose date until the first response CR/PR (maximum duration: 938 days)
  Time to response was defined as the time from first dose date until the first response CR/PR (whichever is first recorded). CR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. PR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters. Time to response was calculated for objective responders only. Confirmation response is required.
Time to Response as per iRECIST | From first dose date until the first response iCR/iPR (maximum duration: 938 days)
  Time to response was defined as the time from first dose date until the first response iCR/iPR (whichever is first recorded). iCR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. iPR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters.Time to response was calculated for objective responders only. Confirmation response is required.

CONTACTS AND LOCATIONS:
Overall Officials: Vice President Medical Sciences - Oncology, Study Director — Astellas Pharma Global Development, Inc.
Locations (54):
- United States (19):
  - Honor Health Research Institute, Scottsdale, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Cancer Center, Fairway, Kansas
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Columbia University Medical Center, New York, New York
  - University Hospital of Cleveland, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Mary Crowley Research Center, Dallas, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (4):
  - Site CA15004, Edmonton, Alberta
  - Site CA15003, Toronto, Ontario
  - Site CA15001, Toronto, Ontario
  - Site CA15002, Montreal, Quebec
- Italy (8):
  - Site IT39004, Ancona
  - Site IT39002, Milan
  - Site IT39003, Milan
  - Site IT39008, Milan
  - Site IT39009, Milan
  - Site IT39010, Modena
  - Site IT39005, Monza
  - Site IT39011, Negrar
- Site JP81001, Chūōku, Japan
- Portugal (2):
  - Site PT35101, Lisbon
  - Site PT35106, Porto
- South Korea (5):
  - Site KR82004, Goyang-si, Gyeonggi-do
  - Site KR82005, Seongnam-si, Gyeonggi-do
  - Site KR82001, Seoul
  - SIte KR82002, Seoul
  - Site KR82006, Seoul
- Spain (8):
  - Site ES34002, Barcelona
  - Site ES34003, Barcelona
  - Site ES34009, Barcelona
  - Site ES34010, Barcelona
  - Site ES34001, Madrid
  - Site ES34006, Madrid
  - Site ES34013, Madrid
  - Site ES34014, Valencia
- Taiwan (3):
  - Site TW88602, Taichung
  - Site TW88601, Tainan
  - Site TW88603, Taipei
- United Kingdom (4):
  - Site GB44003, London
  - Site GB44006, London
  - Site GB44004, Newcastle upon Tyne
  - Site GB44005, Sutton Surry

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/8374-CL-0101/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14563&tenant=MT_AST_9011